CLINICAL TRIAL: NCT04207840
Title: Study of Drug Exposure in Systemic Circulation of Primatene Mist (0.25mg) by Oral Inhalation, Versus Epinephrine Injection (0.30mg) by Intramuscular Injection and ProAir (0.18mg) by Oral Inhalation in Healthy Individuals: A Randomized, Safety Evaluator-blind, Three-Treatment, Crossover, Fasting Study
Brief Title: Study of Drug Exposure in Systemic Circulation of Primatene Mist by Oral Inhalation, Versus Epinephrine Injection by Intramuscular Injection and ProAir by Oral Inhalation in Healthy Individuals
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: API-E004-CL-I
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Results first posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Pharmacokinetics; Epinephrine; Albuterol; Asthma; Anaphylaxis
MeSH Terms: conditions — Asthma; Anaphylaxis | interventions — Epinephrine; Inhalation; Albuterol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Primatene Mist, E004 (Experimental): Participants who dosed with Primatene Mist.
  Interventions: Combination Product: Epinephrine (0.125 mg/inhalation)
- Epinephrine Injection Auto-Injector (Generic of EpiPen) (Active Comparator): Participants who were dosed with an Epinephrine Injection Auto-Injector.
  Interventions: Combination Product: Epinephrine Injection Auto-Injector (0.3mg/0.3mL)
- Albuterol HFA (Active Comparator): Participants who dosed with Albuterol HFA.
  Interventions: Combination Product: Albuterol Sulfate (0.09 mg/inhalation)

INTERVENTIONS:
Combination Product: Epinephrine (0.125 mg/inhalation) — Participants will self-administer 2 inhalations of Epinephrine (0.125 mg/inhalation) for a total dosage of 0.25 mg.
  Other Names: Primatene Mist
  Arms: Primatene Mist, E004
Combination Product: Epinephrine Injection Auto-Injector (0.3mg/0.3mL) — Participants will receive an intramuscular injection of Epinephrine via Auto-Injector (0.30 mg of epinephrine solution in 0.30 mL). The 0.30 mL dose will be given perpendicularly as a single deep intramuscular injection into the anterolateral aspect of the thigh.
  Other Names: Generic of EpiPen
  Arms: Epinephrine Injection Auto-Injector (Generic of EpiPen)
Combination Product: Albuterol Sulfate (0.09 mg/inhalation) — Participants will self-administer 2 inhalations of Albuterol Sulfate (0.09 mg/inhalation) for a total dosage of 0.18 mg.
  Other Names: Albuterol HFA
  Arms: Albuterol HFA

SUMMARY:
To assess the drug exposure profile in systemic circulation of Primatene Mist by inhalation, versus Epinephrine by intramuscular injection, and ProAir HFA by inhalation in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate; understand and sign informed consent;
* Male and female adults, aged 18 to 50 years, inclusive at Screening;
* Generally healthy and medically stable, with no clinically significant abnormalities based on physical examination and laboratory tests as determined by the Investigators;
* Have good venous access;
* Have normal resting blood pressure and normal heart rate (HR) without history of syncope; a subject with out of range blood pressure may be enrolled in the study at the discretion of the Principal Investigator;
* Have a body mass index (BMI) of 18.0 - 30.0 kg/m^2;
* Female candidates must be >1 year post-menopausal or practicing a clinically acceptable form of birth control and confirmed by negative urine or serum pregnancy test at Screening;
* Negative HIV-Ab, HBs-Ag and HCV-Ab;
* Negative alcohol test (urine or breathalyzer);
* Negative drug screening results;
* Currently non-smoker; have not used any tobacco products for at least three (3) months prior to Screening; and
* Demonstrate proficiency in the use of MDI and a consistent inhalation time >2.0 seconds after training, for at least three (3) times, with a maximum of 5 attempts.

Exclusion Criteria:

* Concurrent clinically significant cardiovascular, hematological, renal, neurologic, hepatic, endocrine, psychiatric, or malignant diseases.
* Known intolerance or hypersensitivity to any component of the study drugs (i.e., Epinephrine, Albuterol Sulfate or any sympathomimetic drugs, HFA-134a, thymol, ethanol, ascorbic acid, nitric acid, and hydrochloric acid).
* Upper or lower respiratory tract infection, or other systemic infection within 6 weeks prior to Screening;
* Clinically significant abnormalities in the screening/baseline ECG; prolonged corrected QT interval (QTcF) on ECG: men >450ms, women: >470ms; single or multiple premature ventricular contractions (PVC);
* Abnormal thyroid function test (if TSH is out of range, refer to T3/T4 for thyroid function assessment);
* Subject has been on other investigational drug/device studies within 30 days of Screening Visit or planned participation in another investigational drug trial at any time during this trial;
* Women who are pregnant or lactating or planning a pregnancy during the study period;
* Subject has donated or lost > 500 mL of blood within 3 months of Screening;
* Evidence of alcohol or drug abuse or dependency within 6 months prior to screening; or
* Use of any of the prohibited drugs without appropriate washout.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Amphastar Study Site 0035, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Access to patient level data and supporting clinical documents may be requested by qualified researchers. Requests will be reviewed on the basis of scientific merit. Patient data will be de-identified to protect the privacy of trial patients in line with applicable laws and regulations.

REFERENCES:
- [Derived] Zhang JY, Luo MZ, Marrs T, Kerwin EM, Bukstein DA. Comparison of Systemic Exposure Between Epinephrine Delivered via Metered-Dose Inhalation and Intramuscular Injection. J Aerosol Med Pulm Drug Deliv. 2025 Apr;38(2):71-82. doi: 10.1089/jamp.2024.0025. Epub 2024 Aug 29. PMID 39207239

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to receive all 3 treatments over 3 treatment periods in a crossover design.
Groups:
- A-B-C: Subjects received one of the three treatments during each study visit. Visit 1: Treatment A: Two (2) inhalations of Primatene Mist (0.125 mg of epinephrine per inhalation), for a total dosage of 0.25 mg; Visit 2: Treatment B: Intramuscular injection of Epinephrine via Auto-Injector (0.30 mg of epinephrine solution in 0.30 mL), for a total dosage of 0.30 mg; Visit 3: Treatment C: Two (2) inhalations of Albuterol HFA (0.09 mg of albuterol sulfate per inhalation), for a total dosage of 0.18 mg.
- B-C-A: Subjects received one of the three treatments during each study visit. Visit 1: Treatment B: Intramuscular injection of Epinephrine via Auto-Injector (0.30 mg of epinephrine solution in 0.30 mL), for a total dosage of 0.30 mg; Visit 2: Treatment C: Two (2) inhalations of Albuterol HFA (0.09 mg of albuterol sulfate per inhalation), for a total dosage of 0.18 mg; Visit 3: Treatment A: Two (2) inhalations of Primatene Mist (0.125 mg of epinephrine per inhalation), for a total dosage of 0.25 mg.
- C-A-B: Subjects received one of the three treatments during each study visit. Visit 1: Treatment C: Two (2) inhalations of Albuterol HFA (0.09 mg of albuterol sulfate per inhalation), for a total dosage of 0.18 mg; Visit 2: Treatment A: Two (2) inhalations of Primatene Mist (0.125 mg of epinephrine per inhalation), for a total dosage of 0.25 mg; Visit 3: Treatment B: Intramuscular injection of Epinephrine via Auto-Injector (0.30 mg of epinephrine solution in 0.30 mL), for a total dosage of 0.30 mg.
Period: Treatment Period 1
Arm/Group | A-B-C | B-C-A | C-A-B
Started | 9 | 10 | 9
Completed | 9 | 10 | 9
Not Completed | 0 | 0 | 0
Period: Washout Period 1 (2-7 Days)
Arm/Group | A-B-C | B-C-A | C-A-B
Started | 9 | 10 | 9
Completed | 9 | 10 | 8
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Treatment Period 2
Arm/Group | A-B-C | B-C-A | C-A-B
Started | 9 | 10 | 8
Completed | 9 | 10 | 8
Not Completed | 0 | 0 | 0
Period: Washout Period 2 (2-7 Days)
Arm/Group | A-B-C | B-C-A | C-A-B
Started | 9 | 10 | 8
Completed | 9 | 10 | 7
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Treatment Period 3
Arm/Group | A-B-C | B-C-A | C-A-B
Started | 9 | 10 | 7
Completed | 9 | 10 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All participants who have been randomized.
Arm/Group | All Study Participants
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 13
  Black or African-American | 10
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  American Indian or Alaska Native | 0
  Other | 4

OUTCOME MEASURES:

1. Primary Outcome: C[Max], Maximum Plasma Concentration of Albuterol or Epinephrine
Description: Pharmacokinetic (PK) blood samples will be collected starting 30 minutes before dose and until 24 hours after dose. Plasma will be isolated for analyzing the concentrations of Albuterol and Epinephrine. C[max] will be obtained directly from the plot of PK curve.
Time Frame: Samples were drawn at 30 minutes pre-dose and at 1, 2, 3, 5, 7, 9, 12, 15, 18, 21, 25, 30, 40, 50, 60, 70, 80, 90, 120 minutes, 4, 6, 8, 12, 18, and 24 hours post-dose.
Population: Per Protocol Population, defined as all subjects who have received all study medications and are evaluable for all treatments.
Measure: Geometric Mean (Standard Deviation); unit: pg/mL
Arm/Group | Primatene Mist, E004 | Epinephrine Injection Auto-Injector (Generic of EpiPen) | Albuterol HFA
Number analyzed (Participants) | 24 | 24 | 24
pg/mL | 240.8 (2.4) | 704.8 (1.8) | 599.8 (1.7)

2. Primary Outcome: AUC(0-tm)_TOT, Area Under the Curve (AUC) of Total (Exogenous and Endogenous, if Available) Active Product Ingredient (API) From Time 0 to Time (tm)
Description: Pharmacokinetic (PK) blood samples will be collected starting 30 minutes before dose and until 24 hours after dose. Plasma will be isolated for analyzing the concentrations of Albuterol and Epinephrine. AUC(0-tm)_TOT will be calculated with the trapezoid method. Time tm is defined as the time after C[max] is reached where API concentration is reduced to the levels of the same day baseline.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: pg/mL x hr
Arm/Group | Primatene Mist, E004 | Epinephrine Injection Auto-Injector (Generic of EpiPen) | Albuterol HFA
Number analyzed (Participants) | 24 | 24 | 24
pg/mL x hr | 26.8 (3.1) | 509.9 (1.5) | 3332.3 (1.3)

3. Primary Outcome: AUC(0-tm)_DE, Area Under the Curve (AUC) of Exogenous Active Product Ingredient (API) From Time 0 to Time (tm)
Description: Pharmacokinetic (PK) blood samples will be collected starting 30 minutes before dose and until 24 hours after dose. Plasma will be isolated for analyzing the concentrations of Albuterol and Epinephrine. AUC(0-tm)_DE will be calculated with the trapezoid method. Time tm is defined as the time after C[max] is reached where API concentration is reduced to the levels of the same day baseline.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: pg/mL x hr
Arm/Group | Primatene Mist, E004 | Epinephrine Injection Auto-Injector (Generic of EpiPen) | Albuterol HFA
Number analyzed (Participants) | 24 | 24 | 24
pg/mL x hr | 18.4 (3.6) | 396.3 (1.6) | 3332.3 (1.3)

4. Primary Outcome: AUC(0-inf), Area Under the Curve (AUC) of Albuterol or Epinephrine From Time 0 to Infinity
Description: Pharmacokinetic (PK) blood samples will be collected starting 30 minutes before dose and until 24 hours after dose. Plasma will be isolated for analyzing the concentrations of Albuterol and Epinephrine. AUC(0-inf) will be calculated with the extrapolation method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: pg/mL x hr
Arm/Group | Primatene Mist, E004 | Epinephrine Injection Auto-Injector (Generic of EpiPen) | Albuterol HFA
Number analyzed (Participants) | 24 | 24 | 24
pg/mL x hr | 18.4 (3.6) | 411.4 (1.7) | 3650.4 (1.3)

5. Secondary Outcome: t[Max], Time at Which Maximum Plasma Concentration of Albuterol or Epinephrine is Observed
Description: Pharmacokinetic (PK) blood samples will be collected starting 30 minutes before dose and until 24 hours after dose. Plasma will be isolated for analyzing the concentrations of Albuterol and Epinephrine. t[max] will be obtained directly from the plot of PK curve when the maximum concentration is observed.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: min
Arm/Group | Primatene Mist, E004 | Epinephrine Injection Auto-Injector (Generic of EpiPen) | Albuterol HFA
Number analyzed (Participants) | 24 | 24 | 24
min | 2.6 (3.0) | 8.3 (2.7) | 21.8 (3.1)

6. Secondary Outcome: t[1/2], Terminal Elimination Half-life of Albuterol or Epinephrine
Description: Pharmacokinetic (PK) blood samples will be collected starting 30 minutes before dose and until 24 hours after dose. Plasma will be isolated for analyzing the concentrations of Albuterol and Epinephrine.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: min
Arm/Group | Primatene Mist, E004 | Epinephrine Injection Auto-Injector (Generic of EpiPen) | Albuterol HFA
Number analyzed (Participants) | 24 | 24 | 24
min | 7.1 (5.2) | 138.8 (4.0) | 420.7 (1.2)

ADVERSE EVENTS:
Time Frame: From signing of consent until follow-up (approximately 4 weeks)
Arm/Group | Primatene Mist, E004 | Epinephrine Injection Auto-Injector (Generic of EpiPen) | Albuterol HFA
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/26 | 0/28
Other Adverse Events (participants affected / at risk) | 3/27 | 1/26 | 2/28
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primatene Mist, E004 (N=27) | Epinephrine Injection Auto-Injector (Generic of EpiPen) (N=26) | Albuterol HFA (N=28)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Injection Site Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT04207840/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT04207840/SAP_001.pdf